CLINICAL TRIAL: NCT06146959
Title: Effect of Corrective Calcaneal Kinesiology Tape on Pain, Function and Sonographic Picture of Plantar Fasciitis in Adolescents With Pronated Foot
Brief Title: Corrective Calcaneal Kinesiology Tape in Adolescents With Pronated Foot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Tayseer Saber Abdeldayem, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004632
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Physical Disability; Physical Therapy Modalities
Keywords: Kinesiology tape , plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: will receive corrective kinesiotaping (50-75% stretch) for 4 weeks, 2 times per week, with 1 day rest
  Interventions: Device: Corrective Kinesiology taping
- Group B (Active Comparator): Group B will receive a home program of intrinsic foot strengthening and stretching exercises.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Device: Corrective Kinesiology taping — corrective kinesiology tape is a form of biomechanical tape that is used with specific tension to get a corrective effect
  Other Names: Kinesiotape
  Arms: Group A
Other: Home exercise program — Intrinsic foot strengthening and stretching exercises
  Arms: Group B

SUMMARY:
The aim of this study is to find the effect of a program of corrective kinesiotaping on pain intensity, foot function, and the sonographic picture of plantar fascia in adolescents with pronated feet.This study hypothesizes that there will be a statistically significant effect of a program of application of the corrective technique of kinesiotaping on plantar heel pain, foot function, and the sonographic picture of plantar fascia in a sample of Egyptian adolescents suffering from pronated feet.

DETAILED DESCRIPTION:
This study will be conducted to find the effect of a program of corrective kinesiotaping on pain intensity, foot function, and the sonographic picture of the plantar fascia in adolescents with pronated feet. Thirty adolescents suffering from plantar heel pain associated with pronated feet will be included in this study. They will be distributed randomly into 2 groups: Group A will receive corrective kinesiotaping (50-75% stretch) for 6 weeks, 2 times per week with 1 day of rest; Group B will receive a home program of intrinsic foot strengthening and stretching exercises. Data will be collected pre- and post-intervention for all groups by using the visual analog scale (VAS), the first two subscales of the foot function index (FFI), and a sonographic picture of the foot for each adolescent. Participants will be recruited from outpatient clinics and schools.

ELIGIBILITY:
Inclusion Criteria:

* Children with unilateral or bilateral plantar fasciitis.
* pronated foot or foot on weightbearing in the navicular drops test.
* Pain and tenderness to palpation at the medial tubercle of the calcaneus for a minimum of 6 weeks and maximum of 6 months

Exclusion Criteria:

* Corticosteroid injection of the heel within the past 3 months.
* Posterior heel pain.
* Systemic inflammatory conditions.
* Diabetes.
* Surgery of the foot.
* Neuromuscular conditions e.g. CP.
* Individuals with BMI > 25.
* Individuals engaged in regular athletic activities

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale | 4 weeks
  minimum score is 0, and the maximum score is 10 ; higher scores means worse outcome

SECONDARY OUTCOMES:
Foot function Index | 4 weeks
  This questionnaire has been designed to give therapists information on how foot pain has affected your ability to to manage in everyday life. each question on a scale from 0 (no pain) to 10 (worst pain imaginable)

OTHER OUTCOMES:
Diagnostic ultrasound | 4 weeks
  A sonographic picture of plantar fascia

CONTACTS AND LOCATIONS:
Overall Officials: Tayseer S Abdeldayem, PhD, Principal Investigator — Beni-Suef University
Locations (1):
- Tayseer Younes, Cairo, Cairo Governorate, Egypt